CLINICAL TRIAL: NCT04596709
Title: Investigation of Blood Glucose and Insulin Response After Intake of Vitalose and Isomaltulose in Comparison to Sucrose and Glucose
Brief Title: Investigation of Blood Glucose and Insulin Response After Intake of Vitalose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beneo-Institute (Industry)
Collaborators: BioTeSys GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: BTS1586/20
Record Dates: First submitted 2020-09-28; First posted 2020-10-22 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Healthy Adults
MeSH Terms: interventions — isomaltulose; Sucrose; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitalose (Active Comparator): dissolved in water
  Interventions: Dietary Supplement: Vitalose
- isomaltulose (Active Comparator): dissolved in water
  Interventions: Dietary Supplement: isomaltulose
- sucrose (Placebo Comparator): dissolved in water
  Interventions: Dietary Supplement: sucrose
- glucose (Placebo Comparator): dissolved in water
  Interventions: Dietary Supplement: glucose

INTERVENTIONS:
Dietary Supplement: Vitalose — dissolved in water
  Arms: Vitalose
Dietary Supplement: isomaltulose — dissolved in water
  Arms: isomaltulose
Dietary Supplement: sucrose — dissolved in water
  Arms: sucrose
Dietary Supplement: glucose — dissolved in water
  Arms: glucose

SUMMARY:
The aim of this study is to assess the postprandial glucose and insulin response of Vitalose.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults
* Age 18-50 years
* BMI ≥18.5 and ≤30.0 kg/m²

Exclusion Criteria:

* acute or chronic disease
* food allergy or intolerance
* intake of medications which affect glucose tolerance

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
2h iAUC for pp glucose response | Baseline, 15, 30, 45, 60, 90, 120 minutes
2h iAUC for pp insulin response | Baseline, 15, 30, 45, 60, 90, 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Menzel, Dr., Principal Investigator — BioTeSys GmbH
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: No